CLINICAL TRIAL: NCT02913963
Title: Changes on Pain and Range of Motion by the Use of Kinesio Taping With Its Corrective of Space Variant on Upper Trapezius Muscle in Subjects With Myofascial Trigger Point
Brief Title: Changes on Pain and Range of Motion by the Use of Kinesio Taping in Subjects With Myofascial Trigger Point
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Fco. Javier Montanez Aguilera, PhD, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEU Cardenal H
Record Dates: First submitted 2016-09-18; First posted 2016-09-26 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Mobility Limitation; Myofascial Trigger Point Pain
MeSH Terms: conditions — Mobility Limitation; Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping (Active Comparator): Four Kinesio Taping strips will be placed with tension on skin forming an asterisk. The point of intersection of the four strips will be just above the myofascial trigger point. The subject will remain three days with the strips on his skin
  Interventions: Device: Kinesio Taping
- Sham Kinesio Taping (Placebo Comparator): Four Kinesio Taping strips will be placed without tension on skin forming an asterisk. The point of intersection of the four strips will be just above the myofascial trigger point. The subject will remain three days with the strips on his skin
  Interventions: Device: Sham Kinesio Taping

INTERVENTIONS:
Device: Kinesio Taping — Four Kinesio Taping strips will be placed with tension on skin forming an asterisk. The point of intersection of the four strips will be just above the myofascial trigger point. The subject will remain three days with the strips on his skin
  Arms: Kinesio Taping
Device: Sham Kinesio Taping — Four Kinesio Taping strips will be placed without tension on skin forming an asterisk. The point of intersection of the four strips will be just above the myofascial trigger point. The subject will remain three days with the strips on his skin
  Arms: Sham Kinesio Taping

SUMMARY:
The aim of this study is to demonstrate that the application of Kinesio Taping on a myofascial trigger point in the trapezius muscle able to cause a decrease of the trigger point pain and an increase of the cervical range of motion in asymptomatic subjects

DETAILED DESCRIPTION:
The use of Kinesio Taping has become very popular for the treatment of many musculoskeletal disorders in recent decades. Of the six variants of application that has the Kinesio Taping, the space correction technique is suggested for pain management. The increased space achieved with this variant decreases the pressure Kinesio Taping by raising the skin directly over the treatment area, reducing chemical irritation receptors and therefore pain. The aim of this study is to demonstrate that the application of this variant of Kinesio Taping on a myofascial trigger point in the trapezius muscle able to cause a decrease of the pain and an increase of the cervical range of motion in asymptomatic subjects. For this, the pressure pain threshold will be measured with a algometer on the trigger point and the range of motion with a cervical goniometer.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study (signed informed consent)
* Presence of latent myofascial trigger point in upper trapezius.

Exclusion Criteria:

* Subjects in which not clearly identified myofascial trigger point in the upper trapezius .
* Subjects who suffer or have suffered pathologies of upper limb deformities or orthopedic injuries that can alter static and biomechanics of shoulder and neck.
* Subjects who suffer or have suffered rheumatic or neurological disease or chronic shoulder pain and/or neck
* Subjects diagnosed with fibromyalgia, myelopathy or radiculopathy.
* Subjects suffering from any psychiatric disorder (such as anxiety or depression).
* Subjects who have suffered post-traumatic alteration (whiplash type) or cervical surgery.
* Pregnancy risk of abortion.
* Have used analgesics in the 48 hours before participating in the study
* Subjects presenting any contraindications to the application of Kinesio Taping.
* Know the Kinesio Taping technique applied in the study.
* Be receiving physical therapy for any shoulder or neck pathology.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-10; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Changes in pressure pain threshold | At the beginning, immediately after intervention and at 72 hours
  Is defined as the minimum force applied which induces pain on myofascial trigger point. Pressure will be applied with algometer

SECONDARY OUTCOMES:
Changes in cervical range of motion | At the beginning, immediately after intervention and at 72 hours
  Cervical range of motion is measuring movement around this segment of the spine. Lateral flexion and rotation. Will be measured with a cervical goniometer

CONTACTS AND LOCATIONS:
Overall Officials: F Javier Montañez-Aguilera, PhD, Study Director — CEU Cardenal Herrera University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva Parreira Pdo C, Menezes Costa Lda C, Takahashi R, Hespanhol Junior LC, Motta Silva T, da Luz Junior MA, Pena Costa LO. Do convolutions in Kinesio Taping matter? Comparison of two Kinesio Taping approaches in patients with chronic non-specific low back pain: protocol of a randomised trial. J Physiother. 2013 Mar;59(1):52; discussion 52. doi: 10.1016/S1836-9553(13)70147-4. PMID 23419916
- [Background] Ekiz T, Aslan MD, Ozgirgin N. Effects of Kinesio Tape application to quadriceps muscles on isokinetic muscle strength, gait, and functional parameters in patients with stroke. J Rehabil Res Dev. 2015;52(3):323-31. doi: 10.1682/JRRD.2014.10.0243. PMID 26220179
- [Background] Gusella A, Bettuolo M, Contiero F, Volpe G. Kinesiologic taping and muscular activity: a myofascial hypothesis and a randomised, blinded trial on healthy individuals. J Bodyw Mov Ther. 2014 Jul;18(3):405-11. doi: 10.1016/j.jbmt.2013.11.007. Epub 2013 Nov 8. PMID 25042311
- [Background] Wu WT, Hong CZ, Chou LW. The Kinesio Taping Method for Myofascial Pain Control. Evid Based Complement Alternat Med. 2015;2015:950519. doi: 10.1155/2015/950519. Epub 2015 Jun 21. PMID 26185522
- [Background] Gerwin RD, Shannon S, Hong CZ, Hubbard D, Gevirtz R. Interrater reliability in myofascial trigger point examination. Pain. 1997 Jan;69(1-2):65-73. doi: 10.1016/s0304-3959(96)03248-4. PMID 9060014
- [Background] Akamatsu FE, Ayres BR, Saleh SO, Hojaij F, Andrade M, Hsing WT, Jacomo AL. Trigger points: an anatomical substratum. Biomed Res Int. 2015;2015:623287. doi: 10.1155/2015/623287. Epub 2015 Feb 24. PMID 25811029
- [Background] Vanderweeen L, Oostendorp RA, Vaes P, Duquet W. Pressure algometry in manual therapy. Man Ther. 1996 Dec;1(5):258-265. doi: 10.1054/math.1996.0276. PMID 11440515
- [Background] Walton DM, Levesque L, Payne M, Schick J. Clinical pressure pain threshold testing in neck pain: comparing protocols, responsiveness, and association with psychological variables. Phys Ther. 2014 Jun;94(6):827-37. doi: 10.2522/ptj.20130369. Epub 2014 Feb 20. PMID 24557645